CLINICAL TRIAL: NCT00352885
Title: IL-2 Neuropsychiatric Symptoms: Mechanism and Prevention
Brief Title: Effectiveness of Escitalopram in Preventing or Reducing Depressive Symptoms in People Receiving Interleukin-2 Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrew H Miller, Professor, Emory University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IRB00024759; R01MH071580 (NIH); DATR A3-NSS
Record Dates: First submitted 2006-07-13; First posted 2006-07-17 (Estimated); Results first posted 2014-06-27 (Estimated); Last update posted 2018-09-14 (Actual); Status verified 2018-08

CONDITIONS: Depression
Keywords: Cancer; IL-2 therapy; Antidepressant; Immune system; Neuroendocrine response
MeSH Terms: conditions — Depression; Neoplasms | interventions — Escitalopram; Sugars; Interleukin-2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escitalopram (Experimental): Participants will receive escitalopram and IL-2 treatment
  Interventions: Drug: Escitalopram; Drug: IL-2
- Placebo (Placebo Comparator): Participants will receive placebo and IL-2 treatment
  Interventions: Drug: Placebo; Drug: IL-2

INTERVENTIONS:
Drug: Escitalopram — Participants will begin medication approximately 2 weeks before their first scheduled IL-2 treatment. The dosage for the first week will be 10 mg per day. If 10 mg is well tolerated by the participant, the dosage will be increased to 20 mg per day. The dosage for the remainder of the study will be 20 mg per day.
  Other Names: Lexapro
  Arms: Escitalopram
Drug: Placebo — Participants will begin the placebo approximately 2 weeks before their first scheduled IL-2 treatment. The dosage for the first week will be 1 pill per day, if 1 pill is well tolerated by the participant the dosage will be increased to 2 pills per day. Two pills per day will be the dosage for the reminder of the study.
  Other Names: Sugar pill
  Arms: Placebo
Drug: IL-2 — IL-2 is a 12-week treatment regimen with intravenous (IV) IL-2. There will be one cycle every 3 weeks for a total of four cycles. One cycle is 720,000 units/kg every 8 hours for 5 days.

SUMMARY:
This study will determine the effectiveness of an antidepressant in preventing or reducing depressive symptoms in people with melanoma who are receiving Interleukin-2 (IL-2) treatment.

DETAILED DESCRIPTION:
Melanoma is the most serious type of skin cancer, affecting nearly 54,000 people in the United States each year. Melanomas often develop in pre-existing moles or as new moles on the body. If left untreated, the cancerous cells can spread throughout the body. Fortunately, melanoma can be cured if a person is diagnosed and treated early. Typical treatments include surgery, amputation, chemotherapy, and immunotherapy. Interleukin-2 (IL-2) treatment, a type of immunotherapy, uses the body's immune system to slow or stop the spread of cancer cells to other parts of the body. However, IL-2 treatment is typically associated with severe side effects, including depression, fatigue, and difficulty thinking. This study will evaluate whether escitalopram, an antidepressant, can help improve treatment-related depressive symptoms, reduce stress hormone levels, and increase the number of treatment cycles among people with metastatic melanoma who are receiving IL-2 treatment.

Participation in this double-blind study will last up to 18 weeks and will include 5 to 14 study visits. Participants will complete four 1-week cycles of IL-2 treatment over a 12-week period. Two weeks prior to starting IL-2 treatment, participants will undergo a psychiatric interview; a computerized thinking test; questionnaires; and blood, urine, and saliva collection. Participants will also be randomly assigned to start receiving either escitalopram or placebo for the entire duration of the study. The dosage of escitalopram or placebo will vary depending on the symptom severity of each participant. Immediately prior to IL-2 treatment, participants will undergo preliminary IL-2 procedures, which will include a medical history review, physical exam, and blood collection. These same procedures will occur every day that the participant is in the hospital for IL-2 treatment. Participants will stay in the hospital when receiving all four IL-2 treatment cycles. During these hospital stays, participants will complete repeat questionnaires and computerized tasks. Blood collection will occur at selected times as well. A follow-up visit will occur 4 weeks after the final treatment dose of IL-2.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cancer and beginning Interleukin (IL)-2 treatment
* Willing to use an effective form of birth control throughout the study if sexually active

Exclusion Criteria:

* Diagnosed with major depression or experiencing significant depressive symptoms or a Hamilton Rating Scale-Depression score of 18 or higher
* Brain metastases, history of a brain injury, or seizure disorders
* Meets Diagnostic and Statistical Manual of Mental Disorders (DSM)-IV criteria for substance abuse or dependence within 3 months of study entry
* Suicidal, psychotic, or received psychiatric hospitalization within 12 months of study entry
* Past or current history of schizophrenia or bipolar disorder
* Pregnant or planning on becoming pregnant within 1 to 2 years
* Evidence of untreated or poorly controlled infectious, hormone, heart, blood, kidney, liver, or neurological disease
* Use of antidepressants, glucocorticoids, guanethidine, centrally acting alpha-antagonists, beta-blockers, or anticonvulsants
* Clinically significant eye abnormalities
* A score lower than 28 on the Mini Mental Status Exam (MMSE)
* Prior history of severe adverse events associated with escitalopram or other selective serotonin reuptake inhibitor (SSRI) antidepressants
* Diagnosed with type 1 or type 2 diabetes
* Any condition that might make the participant unsuitable for enrollment or that could interfere with study participation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-10-06 (Actual); Primary Completion 2010-05-17 (Actual); Study Completion 2010-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique L. Musselman, MD,MS, Principal Investigator — Emory University; David Lawson, MD, Study Chair — Emory University; Andrew Miller, MD, Study Chair — Emory University
Locations (1):
- Winship Cancer Institute, Atlanta, Georgia, United States

REFERENCES:
- [Result] Musselman D, Royster EB, Wang M, Long Q, Trimble LM, Mann TK, Graciaa DS, McNutt MD, Auyeung NS, Oliver L, Lawson DH, Miller AH. The impact of escitalopram on IL-2-induced neuroendocrine, immune, and behavioral changes in patients with malignant melanoma: preliminary findings. Neuropsychopharmacology. 2013 Sep;38(10):1921-8. doi: 10.1038/npp.2013.85. Epub 2013 Apr 10. PMID 23575741
- [Derived] Vita G, Compri B, Matcham F, Barbui C, Ostuzzi G. Antidepressants for the treatment of depression in people with cancer. Cochrane Database Syst Rev. 2023 Mar 31;3(3):CD011006. doi: 10.1002/14651858.CD011006.pub4. PMID 36999619
- [Derived] McNutt MD, Liu S, Manatunga A, Royster EB, Raison CL, Woolwine BJ, Demetrashvili MF, Miller AH, Musselman DL. Neurobehavioral effects of interferon-alpha in patients with hepatitis-C: symptom dimensions and responsiveness to paroxetine. Neuropsychopharmacology. 2012 May;37(6):1444-54. doi: 10.1038/npp.2011.330. Epub 2012 Feb 22. PMID 22353759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Winship Cancer Institute in Atlanta, Georgia. Participant enrollment began in October 2006 and all study participation ended in May 2010.
Pre-assignment Details: Of 67 approached about the study, 26 met eligibility criteria and consented to participate in the trial. Two individuals did not come to the screening visit leaving 24 that were randomized evenly between the study arms. An additional 4 participants were discontinued prior to beginning IL-2 therapy, resulting in 20 participants who began the study.
Groups:
- Escitalopram: Participants receiving 10-20 mg of escitalopram per day from two weeks before IL-2 treatment begins and continuing through the duration of IL-2 treatment. IL-2 treatment consists of four 3-week cycles, for 12 weeks of IL-2 treatment and a total of 14 weeks of the escitalopram intervention.
- Placebo: Participants receiving a placebo from two weeks before IL-2 treatment begins and continuing through the duration of IL-2 treatment. IL-2 treatment consists of four 3-week cycles, for 12 weeks of IL-2 treatment and a total of 14 weeks of the intervention of a placebo to match escitalopram.
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 9 | 11
Completed Cycle 1 of IL-2 Treatment | 9 | 11
Completed Cycle 2 of IL-2 Treatment | 8 | 9
Completed Cycle 3 of IL-2 Treatment | 4 | 7
Completed (Completed all four cycles of IL-2 treatment) | 3 | 4
Not Completed | 6 | 7
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Development of major depression | 0 | 1
Not completed — Progression of metastatic melanoma | 5 | 3
Not completed — Side effects of IL-2 administration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (8.4) | 44.6 (16.1) | 47.4 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 7 | 8 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9 | 11 | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of IL-2 Treatments Tolerated
Description: The mean number of IL-2 doses tolerated (out of the possible 60 total doses) are presented for each study arm. The standard high dose regimen of IL-2 includes 15 doses per cycle. The dose of IL-2 is reduced, or treatment is stopped entirely, if the side effects become severe. This analysis includes the total number of doses taken at the end of Cycle 4, by all participants who began the trial, regardless of how many cycles each participant completed.
Time Frame: Cycle 4 (up to 12 weeks of IL-2 treatment)
Measure: Mean (Standard Deviation); unit: IL-2 treatments
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 9 | 11
IL-2 treatments | 18.4 (8.22) | 19.8 (8.96)

2. Secondary Outcome: Plasma Concentrations of Adrenocorticotropic Hormone (ACTH)
Description: Adrenocorticotropic hormone (ACTH) is a stress hormone that is synthesized by the pituitary in response to corticotropin-releasing hormone (CRH). ACTH stimulates adrenal cortisol production. ACTH levels vary throughout the day and are highest between 6am and 8am. A typical reference range is 10-50 picograms per milliliter (pg/ml) from blood drawn in the morning. Low levels of ACTH can indicate adrenal insufficiency (including adrenal cancers) while high levels may indicate several diseases or stress. IL-2 treatment stimulates the release of ACTH and this stimulation is dose dependent (rising as the dose of IL-2 increases) and tends to increase further with repeated exposure to IL-2. Blood was drawn for measuring ACTH at screening (baseline value) and once during days 1-3 of each cycle of the four IL-2 treatments.
Time Frame: Screening and Cycles 1 - 4 (up to 14 weeks)
Population: The population in this analysis includes participants with ACTH measurements at the indicated study visit. Participants withdrew or were terminated from the study early depending on their ability to continue IL-2 treatment.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 9 | 11
pg/ml
  Screening | 27.55 (7.41) | 28.95 (4.43)
  Cycle 1 | 45.66 (7.58) | 56.60 (10.46)
  Cycle 2: number analyzed (Participants) | 8 | 9
  Cycle 2 | 112.59 (73.04) | 75.69 (20.61)
  Cycle 3: number analyzed (Participants) | 4 | 7
  Cycle 3 | 87.89 (36.03) | 136.13 (60.52)
  Cycle 4: number analyzed (Participants) | 3 | 4
  Cycle 4 | 91.25 (45.23) | 81.23 (22.08)

3. Secondary Outcome: Plasma Concentrations of Interleukin 6 (IL-6)
Description: Immune system functioning was assessed by measuring plasma concentrations of interleukin 6 (IL-6). IL-6 is a proinflammatory cytokine that is elevated during times of inflammation, infection, in patients with advanced or metastatic cancer, and is also implicated in mood disorders. IL-2 treatments are associated with increased IL 6 levels, in a dose response manner. IL-6 values in healthy individuals are generally less than 16 pg/ml. Blood was drawn for measuring IL-6 at screening (baseline value) and once during days 1-3 of each cycle of the four IL-2 treatments.
Time Frame: Screening and Cycles 1 - 4 (up to 14 weeks)
Population: The population in this analysis includes participants with IL-6 measurements at the indicated study visit. Participants withdrew or were terminated from the study early depending on their ability to continue IL-2 treatment.
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 9 | 11
pg/ml
  Screening | 11.68 (7.09) | 10.12 (3.36)
  Cycle 1 | 290.77 (81.63) | 270.11 (71.85)
  Cycle 2: number analyzed (Participants) | 8 | 9
  Cycle 2 | 210.90 (49.96) | 297.94 (67.94)
  Cycle 3: number analyzed (Participants) | 4 | 7
  Cycle 3 | 305.41 (69.95) | 332.49 (52.54)
  Cycle 4: number analyzed (Participants) | 3 | 4
  Cycle 4 | 283.34 (67.55) | 308.09 (57.37)

4. Secondary Outcome: Plasma Concentrations of Cortisol
Description: Cortisol is a steroid hormone made in the adrenal glands in response to fear or stressful situations. A typical reference range is 6-23 micrograms/deciliter (mcg/dL) from blood drawn in the morning. Low levels of cortisol can indicate Addison's disease or a problem with the pituitary gland, while high levels may indicate tumors of the adrenal gland, among other illnesses, or increased stress. Chronic elevation of cortisol is associated with reduced immune function and increased risk of heart disease. IL-2 treatment stimulates the release of cortisol and this stimulation is dose dependent (rising as the dose of IL-2 increases) and tends to increase further with repeated exposure to IL-2. Blood was drawn for measuring cortisol at screening (baseline value) and once during days 1-3 of each cycle of the four IL-2 treatments.
Time Frame: Screening and Cycles 1 - 4 (up to 14 weeks)
Population: The population in this analysis includes participants with cortisol measurements at the indicated study visit. Participants withdrew or were terminated from the study early depending on their ability to continue IL-2 treatment.
Measure: Mean (Standard Error); unit: mcg/dL
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 9 | 11
mcg/dL
  Screening | 11.51 (2.06) | 10.62 (1.27)
  Cycle 1 | 20.60 (1.47) | 17.78 (1.58)
  Cycle 2: number analyzed (Participants) | 8 | 9
  Cycle 2 | 19.53 (2.53) | 18.46 (1.79)
  Cycle 3: number analyzed (Participants) | 4 | 7
  Cycle 3 | 22.44 (2.39) | 19.11 (1.15)
  Cycle 4: number analyzed (Participants) | 3 | 4
  Cycle 4 | 20.58 (2.63) | 18.86 (1.29)

5. Secondary Outcome: Hamilton Depression Rating Scale (HAM-D) Score
Description: Hamilton Depression Rating Scale (HAM-D) is a 21-item, observer-rated scale which quantifies the severity of depressive symptoms, including depressed mood, loss of interest in usually pleasurable activities, insomnia, anorexia, fatigue, weight loss, and psychomotor retardation or agitation. Participants rate the severity of their symptoms on a scale of 0-2 or 0-4 (depending on the item), where 0 means that the symptom is absent. Total scores are calculated by summing the first 17 items for a total score between 0 and 50. For this study a score of 0-6 indicates a normal state, a score of 7-17 indicates mild depression, a score of 18-24 indicates moderate depression, and a score of greater than 25 indicates severe depression. The HAM-D was administered at screening (baseline value) and once during days 1-3 of each cycle of the four IL-2 treatments.
Time Frame: Screening and Cycles 1 - 4 (up to 14 weeks)
Population: The population in this analysis includes participants completing the HAM-D at the indicated study visit. Participants withdrew or were terminated from the study early depending on their ability to continue IL-2 treatment.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 9 | 11
units on a scale
  Screening | 7.77 (1.27) | 6.45 (1.51)
  Cycle 1 | 11.56 (2.24) | 12.73 (1.63)
  Cycle 2: number analyzed (Participants) | 8 | 9
  Cycle 2 | 12.33 (1.69) | 15.00 (2.05)
  Cycle 3: number analyzed (Participants) | 4 | 7
  Cycle 3 | 14.56 (1.61) | 16.64 (2.38)
  Cycle 4: number analyzed (Participants) | 3 | 4
  Cycle 4 | 14.56 (1.77) | 16.00 (2.45)

6. Secondary Outcome: Genetic Polymorphisms
Time Frame: Screening and After Cycle 4 (up to 14 weeks)
Population: Genetic polymorphisms were not analyzed due to the small sample size and insufficient funds.
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Data were collected for adverse events from the screening visit through the end of IL-2 treatment (up to 14 weeks).
Description: Due to the nature of the underlying illness and treatment with IL-2, many adverse events were expected in this population. Only unexpected adverse events that occurred while a participant was actively taking part in the study are reported.
Arm/Group | Escitalopram | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/11
Serious Adverse Events (participants affected / at risk) | 5/9 | 3/11
Other Adverse Events (participants affected / at risk) | 1/9 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=9) | Placebo (N=11)
Progression of melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Escitalopram (N=9) | Placebo (N=11)
major depression (Psychiatric disorders) | 0 (0) | 1 (1)
cardiac effect (Cardiac disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Barriers to recruitment included: patient refusal of IL-2 treatment, hesitation to join a placebo-controlled trial or take an antidepressant, depression requiring open-label, antidepressant treatment, reluctance to delay IL-2 treatment for two weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No